CLINICAL TRIAL: NCT00515931
Title: Radiation Therapy as Palliative Treatment of GIST Progressing During or After Tyrosine Kinase Inhibitor Therapy: A Prospective Study
Brief Title: Radiation Therapy as Palliative Treatment of GIST
Acronym: GIST-RT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heikki Joensuu (Other)
Collaborators: Lund University (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor-Investigator, Heikki Joensuu, Professor, University of Helsinki
Organization: University of Helsinki (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIST-RT-2007
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Sarcoma
Keywords: Gastrointestinal stromal tumor; GIST; Sarcoma; Radiation therapy; Radiotherapy
MeSH Terms: conditions — Sarcoma; Gastrointestinal Stromal Tumors | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy (Experimental): GIST patients who have progressing metastases will be treated with radiotherapy.
  Interventions: Radiation: Radiation therapy (external beam photons)

INTERVENTIONS:
Radiation: Radiation therapy (external beam photons) — A cumulative radiation dose of 30 to 40 Gy is administered in 1.8 to 2.0 Gy fractions, 5 fractions per week, to the target lesion(s).
  Other Names: Radiotherapy, fractionated radiation therapy

SUMMARY:
Gastrointestinal stromal tumors (GISTs) are generally considered resistant to radiation, but no prospective trials addressing efficacy and tolerability of radiation therapy have been carried out. Limited clinical experience suggests that selected GIST patients may benefit from palliative radiation therapy. The purpose of this prospective, non-randomized, multicenter study is to evaluate efficacy and safety of palliative radiation therapy in GIST patients who have progressive GIST during or after tyrosine kinase inhibitor therapy.

DETAILED DESCRIPTION:
Radiation therapy planning must be based on computerized tomography (CT). External beam radiation must be used. Both 3D and IMRT plans are acceptable. The cumulative radiation dose may range from 30 to 40 Gy as administered in 1.8 to 2.0 Gy fractions, 5 fractions per week. The dose is specified as defined by the ICRU (International Commission on Radiation Units and Measurements) report 50. Response is evaluated using CT 6 and 12 weeks after irradiation. Adverse effects are evaluated using the Common Terminology Criteria for Adverse Effects (CTCAE)version 3.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified GIST.
* Metastatic or locally advanced, inoperable disease.
* Adequate systemic treatment has been administered.
* One or more growing GIST metastasis present during of after TKI therapy.
* The target lesion(s) is measurable.
* A written informed consent

Exclusion Criteria:

* WHO performance status is 4.
* Estimated life-expectancy less than 3 months.
* Radiation planning target volume greater than 3 dm3.
* Unmeasurable target lesion. Bone and brain metastases are not accepted target lesions.
* Radiation therapy cannot be delivered (e.g. active infection or restlessness.)
* Pregnancy.
* Systemic GIST treatment with unknown efficacy.
* Copies of CT images cannot be sent for central review.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Target tumor response rate | 6 to 12 weeks

SECONDARY OUTCOMES:
Time to progression of irradiated lesions | 6 months
Time to progression of GIST | 6 months
Control of GIST-related symptoms | 6 months
Adverse effects of radiation therapy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, M.D., Ph.D., Principal Investigator — Department of Oncology, Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Joensuu H, Eriksson M, Collan J, Balk MH, Leyvraz S, Montemurro M. Radiotherapy for GIST progressing during or after tyrosine kinase inhibitor therapy: A prospective study. Radiother Oncol. 2015 Aug;116(2):233-8. doi: 10.1016/j.radonc.2015.07.025. Epub 2015 Jul 27. PMID 26228971